CLINICAL TRIAL: NCT04907929
Title: Effectiveness Speech and Cognitive Therapy Implant Pre-cohlear Implantation
Acronym: EPOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20-AOIP-02
Record Dates: First submitted 2021-04-28; First posted 2021-06-01 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Cochlear Implants
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- post-implantation care (Experimental)
  Interventions: Behavioral: targeted speech and cognitive therapy

INTERVENTIONS:
Behavioral: targeted speech and cognitive therapy — One month of targeted speech and cognitive therapy with a speech therapist and with home exercice at home by using a numeric solution

SUMMARY:
It has been shown that in deaf people, cortical reorganisation occurs and can accelerate age-related cognitive decline. Therefore, even though a number of Cochlear Implantation Reference Centres are setting up tests to detect cognitive disorders, these remain global and not very specific to deafness. Similarly, auditory rehabilitation could make cognitive decline reversible and bring about major changes in the cognitive functioning of patients which will be decisive for the effectiveness of speech therapy and the effectiveness of implantation. Indeed, it has been shown that, in the deaf postlingual patient, less neuronal activity in the auditory cortex and a reallocation of the cortical regions dedicated to auditory processing to visual tasks took place. This could subsequently influence the outcome of the cochlear implant. The aim of this study is therefore to evaluate the effectiveness of targeted speech therapy aimed at cognitive reorganisation on post-implant gain.

ELIGIBILITY:
Inclusion Criteria:

* Men or Women ≥ 18 years of age coming for consultation at the implementation centre.
* Subjects who can read and write French.
* Patients who are candidates for cochlear implantation and who have not had any contraindication to the operation following the pre-implant assessment.
* Ability to sign free and informed consent.
* Subjects with a smartphone or laptop that allows access to the application

Exclusion Criteria:

- Physical and cultural factors that may interfere with testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Verbal fluency test | 3 months
  This test consists of giving as many words as possible beginning with the same letter in two minutes (phonological fluencies) and as many words of the same category in two minutes (semantic fluencies). The interest of the study of fluencies is that they allow us to observe both the preferred functioning of patients (semantic vs. phonological) and other components such as working memory and semantic memory. The duration of this test is four minutes.
Grober et Buschke's test | 3 months
  This test assesses verbal memory and is composed of 16 items belonging to 16 different semantic categories. Indicative recall is used to check the efficiency of encoding and to dissociate memory disorders according to their type.
Door test | 3 months
  This test assesses visual-spatial episodic memory. It consists of presenting 24 pictures of doors to the patient. The patient must then recognise each of these doors in the presence of three distractors. It is divided into two parts which differ in terms of difficulty of recognition.
Hospital Anxiety end Depression scale | 3 months
  The HAD scale is an instrument to screen for anxiety and depressive disorders. It consists of 14 items rated from 0 to 3. Seven questions relate to anxiety (total A) and seven others to the depressive dimension.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas GUEVARA, Dr, Study Director — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No